CLINICAL TRIAL: NCT00090194
Title: Evaluation of Immune Globulin Intravenous (Human), 10%, Manufactured by Chromatography Process (IGIV-C, 10%), as an Agent to Reduce Anti-HLA Antibodies and Improve Transplantation Results in Cross Match Positive Living Donor Kidney Allograft Recipients
Brief Title: Improving Transplant Options of Highly Sensitized Recipients Using IGIV-C, 10%
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT IG03
Record Dates: First submitted 2004-08-25; First posted 2004-08-26 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Transplantation; Transplantation, Homologous; HLA Antigens; Autoantibodies; Immunoglobulins, Intravenous; Living Donors; Dose-Response Relationship, Immunologic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Experimental): 0.5 gm/kg at 5 days pre-transplant and 7 days post-transplant
  Interventions: Biological: Immune Globulin Intravenous (Human), 10%
- Middle Dose (Experimental): 1.0 gm/kg at 5 days pre-transplant and 7 days post-transplant
  Interventions: Biological: Immune Globulin Intravenous (Human), 10%
- High Dose (Experimental): 2.0 gm/kg at 5 days pre-transplant and 7 days post-transplant
  Interventions: Biological: Immune Globulin Intravenous (Human), 10%

INTERVENTIONS:
Biological: Immune Globulin Intravenous (Human), 10%

SUMMARY:
The purpose of this study is to determine if IGIV-C, 10% will be effective in converting a donor-recipient crossmatch status from positive to negative. The crossmatch test is used to determine if the donor tissue and recipient tissue are compatible. The study will also evaluate if IGIV-C, 10% will allow successful kidney transplantation in a patient who otherwise would not be able to receive a transplant. Three dose levels of IGIV-C, 10% will be evaluated to determine what dose level is most effective.

DETAILED DESCRIPTION:
Kidney transplantation has emerged as the treatment of choice for patients with end-stage renal disease (ESRD). Preliminary data suggest that IGIV therapy could have significant benefits in modifying allograft rejection episodes, stabilizing long-term allograft function, and reducing ischemia/reperfusion injury.

Qualified patients will have an in-vitro assessment of the ability of IGIV-C, 10% to convert the donor-specific crossmatch (cytotoxic assay) from positive to negative. Those patients with successful in-vitro conversion of the donor-specific crossmatch assay will be randomized to receive IGIV-C, 10% intravenously at a dose of either 2 gm/kg, 1 gm/kg, or 0.5 gm/kg. IGIV-C, 10% will be administered 3 to 5 days prior to planned transplantation and, if transplantation is successful, 7 days post-transplant. If after receiving the IGIV-C infusion the donor-specific crossmatch reveals that cell death has fallen to 20% or less above background, the crossmatch will be considered negative. If after receiving one infusion the crossmatch remains positive, additional IGIV-C infusions may be administered at one-month intervals, up to 4 infusions. A repeat crossmatch must be obtained after each infusion. Patients will be followed for 12 months post-transplant. Concomitant therapy will include a standard immunosuppression regimen of mycophenolate mofetil, tacrolimus, and prednisone following induction therapy with thymoglobulin.

ELIGIBILITY:
Inclusion Criteria for Recipient:

* End-stage renal disease
* No known contraindications for therapy with IGIV-C, 10%
* Have identified a living kidney donor
* Positive crossmatch with the intended donor
* Parent or guardian willing to provide consent, if applicable

Exclusion Criteria for Recipient:

* Pregnant or breastfeeding
* Women of child-bearing age who are not willing or able to practice approved methods of contraception
* HIV infection
* Hepatitis B or hepatitis C infection
* History of positive tuberculin skin test
* Selective IgA deficiency, known anti-IgA antibodies, or history of severe allergy to any part of the clinical trial material
* Have received or will receive multiple organ transplants
* Any licensed or investigational live attenuated vaccine within 2 months of the screening visit
* Patients deemed unable to comply with the protocol
* Heart attack within 1 year of screening
* History of clinically significant thrombotic episodes or active peripheral vascular disease
* Investigational agents within 4 weeks of study entry

Inclusion Criteria for Donor:

* Positive donor-specific crossmatch with the intended recipient
* ECOG performance status 0 or 1
* Excellent health
* Acceptable laboratory parameters
* Compatible blood type
* Normal heart and lung evaluations
* Parent or guardian willing to provide consent, if applicable

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-06; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Monitoring of crossmatch conversion rate after one infusion of IGIV

SECONDARY OUTCOMES:
Graft survival and function
average percentage panel reactive antibodies (PRA) reduction
donor-specific unresponsiveness and allo-responsiveness in ESRD patients
subject survival
safety endpoints, including incidence rates of infection, adverse events, and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Stanley C. Jordan, MD, Study Chair — Department of Pediatrics, Cedars-Sinai Medical Center
Locations (16):
- United States (16):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Good Samaritan Regional Medical Center, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Akalin E, Ames S, Sehgal V, Fotino M, Daly L, Murphy B, Bromberg JS. Intravenous immunoglobulin and thymoglobulin facilitate kidney transplantation in complement-dependent cytotoxicity B-cell and flow cytometry T- or B-cell crossmatch-positive patients. Transplantation. 2003 Nov 27;76(10):1444-7. doi: 10.1097/01.TP.0000084200.40159.EC. PMID 14657683
- [Background] Jordan S, Cunningham-Rundles C, McEwan R. Utility of intravenous immune globulin in kidney transplantation: efficacy, safety, and cost implications. Am J Transplant. 2003 Jun;3(6):653-64. doi: 10.1034/j.1600-6143.2003.00121.x. PMID 12780556
- [Background] Jordan SC, Vo A, Bunnapradist S, Toyoda M, Peng A, Puliyanda D, Kamil E, Tyan D. Intravenous immune globulin treatment inhibits crossmatch positivity and allows for successful transplantation of incompatible organs in living-donor and cadaver recipients. Transplantation. 2003 Aug 27;76(4):631-6. doi: 10.1097/01.TP.0000080685.31697.FC. PMID 12973100
- [Background] Jordan SC, Vo AA, Toyoda M, Tyan D, Nast CC. Post-transplant therapy with high-dose intravenous gammaglobulin: Applications to treatment of antibody-mediated rejection. Pediatr Transplant. 2005 Apr;9(2):155-61. doi: 10.1111/j.1399-3046.2005.00256.x. PMID 15787786
- [Background] Zachary AA, Montgomery RA, Ratner LE, Samaniego-Picota M, Haas M, Kopchaliiska D, Leffell MS. Specific and durable elimination of antibody to donor HLA antigens in renal-transplant patients. Transplantation. 2003 Nov 27;76(10):1519-25. doi: 10.1097/01.TP.0000090868.88895.E0. PMID 14657698
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY356 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY356 — ImmPort study identifier is SDY356
- Available data/document: Study Protocol: SDY356 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY356 — ImmPort study identifier is SDY356
- Available data/document: Study summary, -design, -demographics, -lab tests, -study files: SDY356 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY356 — ImmPort study identifier is SDY356